CLINICAL TRIAL: NCT05123976
Title: A Comparative, Open-label, Randomized, Two-period Bioequivalence Study of Olanzapine Film-coated Tablets 5 mg (JSC Farmak, Ukraine) vs Zyprexa® Coated Tablets 5 mg (Eli Lilly, Nederland B V) in Healthy Subjects Under Fasted Conditions.
Brief Title: Fasted Bioequivalence Study of 2 Olanzapine Film-coated Tablets, 5 mg, in Healthy, Adult Male and Female Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joint Stock Company "Farmak" (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FK/ONZP/2019
Record Dates: First submitted 2021-11-15; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Pharmacokinetics
Keywords: bioequivalence; pharmacokinetics; generic drugs; Olanzapine
MeSH Terms: interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Olanzapine film-coated tablets 5 mg (JSC Farmak, Ukraine)
  Interventions: Drug: Olanzapine film-coated tablets 5 mg (JSC Farmak, Ukraine)
- Treatment B (Active Comparator): Zyprexa® coated tablets 5 mg (Eli Lilly, Nederland B V)
  Interventions: Drug: Zyprexa® coated tablets 5 mg (Eli Lilly, Nederland B V)

INTERVENTIONS:
Drug: Olanzapine film-coated tablets 5 mg (JSC Farmak, Ukraine) — After an overnight fast of at least 10 hours, a 1 film-coated tablet was administered orally with 240 mL of water .
  Other Names: Adagio film-coated tablets 5 mg (JSC Farmak, Ukraine)
  Arms: Treatment A
Drug: Zyprexa® coated tablets 5 mg (Eli Lilly, Nederland B V) — After an overnight fast of at least 10 hours, a 1 film-coated tablet was administered orally with 240 mL of water .
  Other Names: Olanzapine
  Arms: Treatment B

SUMMARY:
This study was designed to assess the bioequivalence of Olanzapine tablets of two different manufacturers and to investigate the safety and tolerability of Olanzapine tablets of two different manufacturers.

DETAILED DESCRIPTION:
A comparative, open-label, randomized, two-period, two-treatment, two-sequence, two-way crossover clinical trial to evaluate the bioequivalence of single doses of test product Olanzapine film-coated tablets 5 mg (JSC Farmak, Ukraine) and reference product Zyprexa® coated tablets 5 mg (Eli Lilly, Nederland B V) in healthy, adult male and female subjects under fasted conditions.

During each period 22 blood samples were taken in each Study Period: prior to dosing (-1.0) and 1.0, 2.0, 3.0, 4.0, 4.5, 5.0, 5.5, 6.0, 6.5, 7.0, 7.5, 8.0, 8.5, 9.0, 10.0, 12.0, 14.0, 16.0, 24.0, 48.0 and 72.0 hours after IMP administration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and non-pregnant and no breast-feeding females ), ≥18 and ≤55 years of age ) (on the day of Informed Consent). Caucasian race.
2. Non-smoker or past-smoker (who has stopped smoking at least 6 months before the first dosing).
3. Body Mass Index (BMI) 18.5 to 30.0 kg/m2, inclusive and body weight between 50 kg and 100 kg (on the day of screening).
4. Subject was available for the whole study and has provided his/her written informed consent.
5. Subjects in good health, as determined by screening medical history, physical examination, vital signs assessments (pulse rate, systolic and diastolic blood pressure, and body temperature) and 12-lead ECG. Minor deviations outside the reference ranges were acceptable, if deemed not clinically significant by the Investigator.
6. All laboratory screening results within the normal range. Minor deviations outside the reference ranges were acceptable, if deemed not clinically significant by the Clinical Investigator.
7. Acceptance of use of contraceptive measures during the whole study by both female and male subjects ).

Exclusion Criteria:

1. Gastrontestinal, renal or hepatic diseases and/or pathological findings present or in history, which might interfere with the drug pharmacokinetics. Any pre-existing disease or condition (e.g. hemicolectomy) for which it can be assumed that absorption, distribution, metabolism and excretion of the IMP will be affected.
2. An unusual diet, for whatever reason (e.g. low-sodium), for four weeks prior to receiving the study drug. In any such case subject selection was at the discretion of the Principal Investigator.
3. History, presence or known risk of narrow-angle glaucoma.
4. Acute or chronic diseases and/or clinical finding which may interfere with the aims of the study or with the drug's safety, tolerability, bioavailability and/or pharmacokinetics of the IMP.
5. Previous liver disease or elevations in serum transaminases ALT or AST ≥ 1.0 ULN at the screening.
6. History of kidney disease and with impaired renal function.
7. Known hypersensitivity or idiosyncratic reaction to olanzapine or to any of its excipients or any drug or any substance.
8. Hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption.
9. Any history or presence of asthma (including aspirin-induced asthma) or nasal polyp or NSAII induced urticaria.
10. Presence of out-of-range cardiac interval on the ECG at screening or other clinically significant abnormalities, unless deemed non-significant by the Investigator.
11. Clinically significant illness within 28 days before the first dosing, including major surgery.
12. Any significant clinical abnormality, including a positive result of HBsAg and/or HCV and/or HIV test during screening procedure.
13. Positive result of blood pregnancy test at screening or positive urine pregnancy test at check-in or breast-feeding or lack of results of pregnancy test.
14. Positive results of drugs in urine at screening and at check-in.
15. Positive result of alcohol breath test at screening and at check-in.
16. Positive result of urine cotinine test at screening.
17. Serious mental disease and/or inability to cooperate with clinical team.
18. Sitting blood pressure after a minimum of 5 minutes of rest is out of the range of 90-140 mmHg for systolic BP and/or 60-90 mmHg for diastolic BP and/or heart rate out of the range of 50-100 bpm during the screening procedure.
19. Body ear temperature is out of the range of 35.7-37.6° C at screening and at check-in.
20. Orthostatic hypotension during the screening procedure.
21. Drug, alcohol (of ≥ 40 g per day pure ethanol), solvents or caffeine abuse.
22. Use of organ-toxic drugs or systemic drugs known to substantially alter liver metabolism within 90 days before the first dosing.
23. Use of any prescription medication for a period of 28 days before the first dosing.
24. Use of any OTC (over-the-counter) medication including vitamins, herbal medications and food supplements less than 14 days before the first dosing.
25. Getting a tattoo, body piercing or any cosmetic treatment involving skin piercing within 90 days before the screening unless evaluated by Investigator as non-significant for inclusion in the study.
26. Donation or loss of at least 500 mL of blood within 90 days or donation of plasma or platelets within 14 days before the first dosing.
27. Subjects who have any clinically significant abnormal laboratory safety findings (upon repeat testing, 1 repeat assessment is acceptable) previously or at screening.

    1. Anaemia (haemoglobin below 120 g/L for women and 130 g/L for men)
    2. Leukopenia (value of WBC below 4.00*10_9/L) and/or neutrophilopenia (value of NEU below 2.0 *10 9/L
    3. Thrombocytopenia (value of platelets below 150*10_9/L).
28. Less thay 30 days between exit procedure in previous study and the first dosing in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
AUC(0-72h) | up to 72 hours post-administration
  The area under the plasma concentration-time curve from time zero to sampling time 72 hours calculated by linear trapezoidal rule
Cmax | up to 72 hours post-administration
  Maximum plasma concentration observed.

SECONDARY OUTCOMES:
tmax. | up to 72 hours post-administration
  The time of the maximum plasma drug concentration

CONTACTS AND LOCATIONS:
Overall Officials: Vlad Udovytskyi, Study Chair — Joint Stock Company "Farmak"
Locations (1):
- QUINTA-ANALYTICA s.r.o., Prague, Czechia